CLINICAL TRIAL: NCT06854172
Title: Investigating the Effects of Mindfulness-Based Self-Compassion Training Given to Parents of Children With Cerebral Palsy on Parents' Self-Efficacy, Caregiver Burden, and Emotion Regulation
Status: Active, not recruiting | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Suheyla YURT, PhD student, Ataturk University
Other Study IDs: B.30.2.ATA.0.01.00/436
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-01

CONDITIONS: It is Planned to Provide Self-compassion Training to Parents of Children With Cerebral Palsy
Keywords: mındfulness; self compassion; education; cerebral palsy; parent; care burden; emotional regulation
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Self-compassion training will be given to the experimental group: Awareness-based self-compassion training will be provided to parents of children with cerebral palsy.
  Interventions: Behavioral: Mindfulness based self-compassion training
- The control group will not receive self-compassion training: A control group of parents of children with cerebral palsy who were not given mindfulness-based self-compassion training

INTERVENTIONS:
Behavioral: Mindfulness based self-compassion training — Self-compassion training is a program that aims to help individuals develop a kind, understanding and tolerant approach towards themselves. In this training, individuals learn to be more compassionate towards themselves and to share. This training can help manage negative emotional states such as stress, anxiety and stress and can lead to a healthier internal balance. When combined with mindfulness techniques, self-compassion training allows individuals to accept the moment and develop a more compassionate approach towards themselves. It is thought that this training will be applied to the experimental group to develop parents' feelings of self-compassion and positively affect the parameters of caregiver burden, self-efficacy and emotion regulation designed in the study.
  Groups: Self-compassion training will be given to the experimental group

SUMMARY:
The purpose of this observational study is to learn the effects of Mindfulness-Based Self-Compassion Training given to parents of children with Cerebral Palsy. The main question it aims to answer is:

-Is Mindfulness-Based Self-Compassion Training effective on parents' caregiver burden, self-efficacy, and emotion regulation? Parents who receive self-compassion training will answer survey questions before and after the training.

ELIGIBILITY:
Inclusion Criteria(For parents):

* Having a child diagnosed with cerebral palsy between the ages of 1-18,
* Being literate,
* Not having communication problems,
* Being between the ages of 18-65.

Inclusion Criteria(For childs):

* Having been diagnosed with Cerebral Palsy,
* Being registered in a special education and rehabilitation center.

Exclusion Criteria:

* Caring for other dependents (elderly, disabled, etc.),
* Having a mental illness (major depression, psychosis, etc.),
* Having communication problems,
* Not continuing education.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The universe of the study consists of Special Education and Rehabilitation Centers in Siirt province. There are a total of 3000 patients registered in Special Education and Rehabilitation Centers. The number of children with cerebral palsy is 252. The parents of children who meet the inclusion criteria will be included in the sample of the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
A personal information form will be filled out regarding the descriptive information of the parents in the experimental and control groups. (Personal information form) | Day 1 and up to study completion, average 9 weeks".
  The diagnostic form to be used in collecting research data was created by the researcher in line with the relevant literature. The Personal Information Form includes questions to determine the socio-demographic status of the parents.
A self-efficacy scale will be applied to determine the self-efficacy levels of parents. (Parent self-efficacy scale) | Day 1 and up to study completion, average 9 weeks
  This scale, developed by Guimond et al. and adapted to Turkish by Diken, is an assessment tool for measuring mothers' and fathers' perceptions of self-efficacy in parenting. The scale consists of 17 items in total and is based on a seven-point Likert-type rating system. Parents respond to statements indicating their perceptions of self-efficacy by marking the appropriate option from the following: (1) "Strongly Disagree", (2) "Disagree", (3) "Partially Disagree", (4) "Undecided", (5) "Partially Agree", (6) "Agree", (7) "Strongly Agree". The lowest and highest scores that can be obtained from this scale are 17 and 119, respectively. As the score increases, the positive increase in parents' perceptions of self-efficacy becomes more apparent.
With this scale, the care burden of parents will be evaluated. (Zarit caregiver load scale) | Day 1 and up to study completion, average 9 weeks
  The Zarit Caregiver Burden Scale was initially developed in 1980 to assess the difficulties faced by caregivers of patients with dementia. Later, the scale was also used to evaluate the challenges faced by caregivers of individuals with schizophrenia. The Turkish version of the scale was translated by Özlü and colleagues, and a validity and reliability study was conducted with the relatives of patients with schizophrenia.
  The Turkish version consists of 19 items and is structured around five sub-dimensions: psychological distress, disruption of personal life, irritability and restriction, social relationship deterioration, financial burden, and dependency. These sub-dimensions help to assess the various difficulties experienced by caregivers in more detail. The scale is rated on a Likert-type scale with responses ranging from "never," "rarely," "sometimes," "often," to "almost always," with scores ranging from 1 to 5.
  The Zarit Caregiver Burden Scale is very useful in determining th
In the study, the Cognitive Emotion Regulation Scale will be used to determine parents' emotion regulation. (Cognitive Emotion Regulation Scale) | Day 1 and up to study completion, average 9 weeks
  This scale was developed to measure the emotion regulation skills of adults. A statistically significant relationship (r=-572) was obtained between the Cognitive Emotion Regulation Scale and the Negative Emotion Scale. Cronbach Alpha, item-total, item-remaining, item discrimination and test-retest methods were used within the scope of reliability studies. It was observed that the item-total correlation values of the scale varied between '.188' and '.468', and the item-remaining correlation values varied between '.104' and '.392'. As a result of the item discrimination analysis, it was concluded that each item had a high discrimination feature. The scale has nine sub-dimensions. These are:
  1. Self-blame
  2. Acceptance
  3. Focus on thought
  4. Positive refocusing
  5. Refocusing on plan
  6. Positive reconsideration
  7. Putting into perspective
  8. Catastrophizing
  9. Blaming others

CONTACTS AND LOCATIONS:
Overall Officials: Suheyla Yurt, PhD Student, Principal Investigator — Siirt University; Sibel ASİ KARAKAŞ, Professor, Study Director — Ataturk University
Locations (1):
- Special Education and Rehabilitation Centers, Siirt, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prest KR, Borek AJ, Boylan AR. Play-based groups for children with cerebral palsy and their parents: A qualitative interview study about the impact on mothers' well-being. Child Care Health Dev. 2022 Jul;48(4):578-587. doi: 10.1111/cch.12962. Epub 2022 Feb 1. PMID 35023213
- [Background] van der Kemp J, Ketelaar M, Rentinck ICM, Sommers-Spijkerman MPJ, Benders MJNL, Gorter JW. Exploring Parents' Experiences and Needs During Disclosure of a Cerebral Palsy Diagnosis of Their Young Child: A Scoping Review. Child Care Health Dev. 2024 Nov;50(6):e13327. doi: 10.1111/cch.13327. PMID 39343726
- [Background] Schuling R, Huijbers MJ, van Ravesteijn H, Donders R, Cillessen L, Kuyken W, Speckens AEM. Recovery from recurrent depression: Randomized controlled trial of the efficacy of mindfulness-based compassionate living compared with treatment-as-usual on depressive symptoms and its consolidation at longer term follow-up. J Affect Disord. 2020 Aug 1;273:265-273. doi: 10.1016/j.jad.2020.03.182. Epub 2020 May 4. PMID 32421612